CLINICAL TRIAL: NCT04542720
Title: Decompression Versus Decompression and Fusion for Lumbar Adjacent Segment Disease
Brief Title: Decompression Versus Decompression and Fusion
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Daniel G.Tobert, M.D., Principle Investigator, Massachusetts General Hospital
Other Study IDs: 2020P000603
Record Dates: First submitted 2020-08-27; First posted 2020-09-09 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Adjacent Segment Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observational: Decompression: Eligible patients may have a preference for the surgical procedure they wish to have. In these instances, they may choose to undergo a decompression alone or a decompression with extension of fusion. These patients are eligible for the study and will be enrolled under observational arms. This arm refers to the decompression alone observational study arm.
  Interventions: Procedure: Observational: Decompression
- Observational: Extension Fusion: Eligible patients may have a preference for the surgical procedure they wish to have. In these instances, they may choose to undergo a decompression alone or a decompression with extension of fusion. These patients are eligible for the study and will be enrolled under observational arms. This arm refers to the decompression with extension of fusion observational study arm.
  Interventions: Procedure: Observational: Extension Fusion

INTERVENTIONS:
Procedure: Observational: Decompression — Patients will undergo decompression alone of the supradjacent level. The surgical technique will be surgeon dependent. All surgeons will be encouraged to avoid damaging facet joints above the fusion mass, retaining 50% of the pars of the decompressed level and performing as minimal of a medial facetectomy as necessary.
  Groups: Observational: Decompression
Procedure: Observational: Extension Fusion — Patients will undergo decompression and extension of posterior instrumentation and fusion. This may or may not include exchange of pre-existing instrumentation. The use of interbody cages will be left to the discretion of the treating surgeon. The purpose of introducing this heterogeneity is to increase the generalizability of the trial results. The fusion cohort will not utilize bone morphogenetic protein products.
  Groups: Observational: Extension Fusion

SUMMARY:
Adjacent segment disease (ASD) in the lumbar spine is a well-known sequela of lumbar fusion surgery. The annual incidence of adjacent level re-operation is approximately 3% with a ten-year prevalence of 20-30%. Frequently, the surgical treatment involves decompression of the adjacent level coupled with extension of the instrumentation and fusion. Advocates of this paradigm cite the altered kinematics and biomechanics of levels adjacent to a lumbar fusion mass. Furthermore, decompressed levels adjacent to a fused segments are associated with higher rates of ASD in retrospective studies. Yet, a retrospective review of higher quality data concluded decompression adjacent to single-level fusion provides similar outcomes compared to fusions extending across the decompressed segments.

Given the conflicting data currently available, higher quality data are needed to guide surgical decision-making in ASD. The purpose of this trial is to prospectively compare decompression and decompression with fusion in patients with lumbar ASD.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients at least one year removed from a previous instrumented posterior lumbar fusion
* Patients with any prior posterior fusion involving L2 to the sacrum, whether single-level or multilevel
* Patients with symptoms related to central and lateral recess at the supradjacent level that have persisted despite at least six weeks of non-operative therapy modalities

Exclusion Criteria:

* Patients with previous uninstrumented lumbar fusions
* Patients with traumatic, neoplastic, or infectious etiologies at the adjacent segment
* Patients with prior iliac or sacroiliac fixation and those with nonunion as the primary indication for surgery
* Patients with pre-existing instability at the supradjacent level. The definition of instability will be determined based on standing lateral, flexion and extension plain radiographs. Patients with >3mm of change between these views will be excluded.
* Retrolisthesis will not be a criterion for exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients at least one year removed from a previous instrumented posterior lumbar fusion will be considered for inclusion in this trial. Any prior posterior fusion involving L2 to the sacrum will be included, whether single-level or multilevel. Patients with symptoms related to central and lateral recess at the suprajacent level that have persisted despite at least six weeks of non-operative therapy modalities will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Global Health, Physical | 3 months, 6 months, 1 year, and 2 years post-operation
  Scored by Patient-Reported Outcomes Measurement Information System (PROMIS): 16-68 (higher score = better outcome)
Physical Function, short form 10a (SF10a) | 3 months, 6 months, 1 year, and 2 years post-operation
  Scored by Patient-Reported Outcomes Measurement Information System (PROMIS): 0-62 (higher score = better outcome)

SECONDARY OUTCOMES:
Global Health, Mental | 3 months, 6 months, 1 year, and 2 years post-operation
  Scored by Patient-Reported Outcomes Measurement Information System (PROMIS): 21-68 (higher score = better outcome)
Pain intensity, short form 3a (SF3a) | 3 months, 6 months, 1 year, and 2 years post-operation
  Scored by Patient-Reported Outcomes Measurement Information System (PROMIS): 30-72 (higher score = better outcome)
Anxiety, short form 4a (SF4a) | 3 months, 6 months, 1 year, and 2 years post-operation
  Scored by Patient-Reported Outcomes Measurement Information System (PROMIS): 40-82 (higher score = better outcome)
Depression, short form 4a (SF4a) | 3 months, 6 months, 1 year, and 2 years post-operation
  Scored by Patient-Reported Outcomes Measurement Information System (PROMIS): 41-80 (higher score = better outcome)
Pain interference, short form 4a (SF4a) | 3 months, 6 months, 1 year, and 2 years post-operation
  Scored by Patient-Reported Outcomes Measurement Information System (PROMIS): 41-76 (higher score = better outcome)
Post-operative complication | 3 months, 6 months, 1 year, and 2 years post-operation
  Scored by Clavien-Dindo classification (Grade I, II, IIIa, IIIb, IVa, IVb, and V) defined at https://www.assessurgery.com/clavien-dindo-classification/
Hospital length of stay | 3 months, 6 months, 1 year, and 2 years post-operation
  Scored by how long the patient is in the hospital after operation.
Post-operative narcotic utilization | 3 months, 6 months, 1 year, and 2 years post-operation
  Scored by morphine milligram equivalents (MME) utilized more than 90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Tobert, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sears WR, Sergides IG, Kazemi N, Smith M, White GJ, Osburg B. Incidence and prevalence of surgery at segments adjacent to a previous posterior lumbar arthrodesis. Spine J. 2011 Jan;11(1):11-20. doi: 10.1016/j.spinee.2010.09.026. PMID 21168094
- [Background] Ghiselli G, Wang JC, Bhatia NN, Hsu WK, Dawson EG. Adjacent segment degeneration in the lumbar spine. J Bone Joint Surg Am. 2004 Jul;86(7):1497-503. doi: 10.2106/00004623-200407000-00020. PMID 15252099
- [Background] Lee CK, Langrana NA. Lumbosacral spinal fusion. A biomechanical study. Spine (Phila Pa 1976). 1984 Sep;9(6):574-81. doi: 10.1097/00007632-198409000-00007. PMID 6495027
- [Background] Radcliff KE, Kepler CK, Jakoi A, Sidhu GS, Rihn J, Vaccaro AR, Albert TJ, Hilibrand AS. Adjacent segment disease in the lumbar spine following different treatment interventions. Spine J. 2013 Oct;13(10):1339-49. doi: 10.1016/j.spinee.2013.03.020. Epub 2013 Jun 15. PMID 23773433
- [Background] Maragkos GA, Motiei-Langroudi R, Filippidis AS, Glazer PA, Papavassiliou E. Factors Predictive of Adjacent Segment Disease After Lumbar Spinal Fusion. World Neurosurg. 2020 Jan;133:e690-e694. doi: 10.1016/j.wneu.2019.09.112. Epub 2019 Sep 27. PMID 31568911
- [Background] Smorgick Y, Park DK, Baker KC, Lurie JD, Tosteson TD, Zhao W, Herkowitz HN, Fischgrund JS, Weinstein JN. Single- versus multilevel fusion for single-level degenerative spondylolisthesis and multilevel lumbar stenosis: four-year results of the spine patient outcomes research trial. Spine (Phila Pa 1976). 2013 May 1;38(10):797-805. doi: 10.1097/BRS.0b013e31827db30f. PMID 23169068
- [Background] Dawson L, Zarin DA, Emanuel EJ, Friedman LM, Chaudhari B, Goodman SN. Considering usual medical care in clinical trial design. PLoS Med. 2009 Sep;6(9):e1000111. doi: 10.1371/journal.pmed.1000111. Epub 2009 Sep 29. PMID 19787044